CLINICAL TRIAL: NCT05649982
Title: Optimization of Guidance in a Digital Tool for Problematic Alcohol Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Martin Kraepelien, Licensed clinical psychologist, Principal investigator, PhD, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ALCOHOLDIARY2
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Drinking Excessive

STUDY DESIGN:
Intervention Model Description: 2*2 factorial experiment
Masking Description: The level of added guidance received will be open to the participants. The main outcome of Alcohol consumption will be self-rated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Digital Tool for Problematic Alcohol Use (Experimental): This is the base version of the intervention with no added guidance.
  Interventions: Behavioral: ALVA
- Digital Tool for Problematic Alcohol Use + Extra Telephone Interview (Experimental): This is the same intervention as the base version, with an added mid-treatment telephone interview.
  Interventions: Behavioral: ALVA
- Digital Tool for Problematic Alcohol Use + Written Guidance (Experimental): This is the same intervention as the base version, with added weekly written guidance.
  Interventions: Behavioral: ALVA
- Digital Tool for Problematic Alcohol Use + Extra Telephone Interview and Written Guidance (Experimental): This is the same intervention as the base version, with added weekly written guidance and an added mid-treatment telephone interview.
  Interventions: Behavioral: ALVA

INTERVENTIONS:
Behavioral: ALVA — Behavioural digital self-help intervention

SUMMARY:
The purpose of the study is to evaluate the effects on alcohol consumption, and the consumption of time spent by a qualified clinician, by adding different forms of guidance to a digital intervention based on an alcohol diary and techniques from cognitive behavioral therapy and relapse prevention. The participants will be adults with problematic alcohol use. The trial will be a 2*2 factorial experiment where written guidance and/or an extra mid-treatment telephone interview will be added to the basic digital intervention, by randomization. The randomized factorial experiment will create four equally large groups (1:1:1:1) who will receive different combinations of added guidance. Main outcome will be effects on alcohol consumption. Effects on alcohol consumption will also be combined with clinician time spent on guidance to assess the resource-effectiveness of added forms of guidance.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Access to internet
3. ≥8 points for men and ≥6 points for women on Alcohol Use Disorders Identification Test (AUDIT)

Exclusion Criteria:

1. Insufficient knowledge of the Swedish language
2. Difficulties reading or writing related to a digital intervention.
3. Other ongoing psychological treatment with a content similar to that in the current study (problematic alcohol use).
4. High suicide risk based on telephone assessment.
5. Other urgent need for more intensive psychiatric care, or addiction care services, based on telephone assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Standardized drinks per week (based on Time Line Follow Back) | Immediately after the intervention
  Changes in standardized drinks per week (using Time Line Follow Back)

SECONDARY OUTCOMES:
Standardized drinks per week (based on Time Line Follow Back) | 12 months after intervention
  Changes in standardized drinks per week (using Time Line Follow Back)
Diagnostic criteria Alcohol Use Disorder | 6 months after intervention
  Using SCID-5, number of diagnostic criteria 0-11, lower is better
Credibility/Expectancy questionnaire | Mid-intervention (4 weeks after intervention start)
  Credibility/Expectancy questionnaire, score range 0-50, higher is better
Alcohol Use Disorders Identification Test | 12 months after intervention
  Alcohol Use Disorders Identification Test (AUDIT), score range 0-40, lower is better
Brunnsviken Brief Quality of Life Scale | 12 months after intervention
  Brunnsviken Brief Quality of Life Scale (BBQ), score range 0-96, higher is better
Penn Alcohol Craving Scale | 12 months after intervention
  Penn Alcohol Craving Scale (PACS), score range 0-30, lower is better
Patient Health Questionnaire 9 | 12 months after intervention
  Patient Health Questionnaire 9 (PHQ-9), score range 0-27, lower is better
Generalized Anxiety Disorder 7 | 12 months after intervention
  Generalized Anxiety Disorder 7 (GAD-7), score range 0-21, lower is better
Readiness to change questionnaire | 12 months after intervention
  Readiness to change questionnaire (RCQ), determines if the participant are in a precontemplation phase, contemplation phase or action phase

OTHER OUTCOMES:
Clinician time | Immediately after the intervention
  Time in minutes the clinician spends on the participant giving guidance through telephone calls and/or written guidance, in minutes, lower is better.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Psychiatry Research, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IPD available anonymized on reasonable request.

REFERENCES:
- [Derived] Sundstrom C, Ivanova E, Lindner P, Johansson M, Kraepelien M. Investigating the added effects of guidance in digital psychological self-care for alcohol problems (ALVA)-protocol for a randomized factorial optimization trial. Trials. 2024 Feb 21;25(1):136. doi: 10.1186/s13063-024-07981-6. PMID 38383426